CLINICAL TRIAL: NCT01375218
Title: Efficacy and Satisfaction Comparing Two Braces in the Treatment of DDH in Infants: A Randomized Clinical Trial
Brief Title: Efficacy and Satisfaction Comparing Two Braces in the Treatment of Developmental Dysplasia of the Hip (DDH) in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041101A
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2013-12

CONDITIONS: Hip Dislocation, Congenital; Congenital Deformity of Hip Joint
MeSH Terms: conditions — Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plastizote Brace (Active Comparator)
  Interventions: Other: Plastizote Brace
- Pavlik Brace (Active Comparator)
  Interventions: Other: Pavlik Brace

INTERVENTIONS:
Other: Pavlik Brace — Pavlik Brace
  Arms: Pavlik Brace
Other: Plastizote Brace — Plastizote Brace
  Arms: Plastizote Brace

SUMMARY:
The purpose of this study is to 1) evaluate the effectiveness of the Plastizote abduction brace compared to the Pavlik harness in the treatment of developmental dysplasia of the hip (DDH) and 2) compare parent/caregiver satisfaction between the Plastizote abduction brace and the Pavlik harness. The investigators hope to learn which brace treatment is best for a definable population so the appropriate brace can be chosen initially avoiding the time, expense, and frustration of a failed technique.

ELIGIBILITY:
Inclusion Criteria:

1. 0-2 months of age
2. Nonterratological developmental dysplasia of the hip diagnosed by physical exam and standard of care ultrasound

Exclusion Criteria:

1. Ages greater than 2 months
2. Neurological condition
3. Terratological congenital dysplasia of the hip diagnosed by physical exam and standard of care ultrasound
4. Chromosomal abnormality

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Resolution of instability | 3-4 week interval
  Negative Barlow and Ortolani tests as well as improvement/normalization in ultrasound measured alpha angle and femoral head coverage

SECONDARY OUTCOMES:
Resolution of instability | 6 month interval
  Negative Barlow and Ortolani tests as well as improvement/normalization in ultrasound measured alpha angle and femoral head coverage

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina Research Institute, OrthoCarolina, P.A., Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Dwan K, Kirkham J, Paton RW, Morley E, Newton AW, Perry DC. Splinting for the non-operative management of developmental dysplasia of the hip (DDH) in children under six months of age. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD012717. doi: 10.1002/14651858.CD012717.pub2. PMID 36214650